CLINICAL TRIAL: NCT03779464
Title: Phase II Study of Gemcitabine Plus Nab-paclitaxel Versus S1 Plus Nab-paclitaxel in Metastatic Adenocarcinoma of the Pancreas
Brief Title: Study of Gemcitabine Plus Nab-paclitaxel Versus S1 Plus Nab-paclitaxel in Metastatic Adenocarcinoma of the Pancreas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of Gastrointestinal Oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHZL-001
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer; Nab-paclitaxel; Gemcitabine; S1
Keywords: pancreatic cancer; nab-paclitaxel; gemcitabine; S1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S/nab (Experimental): Nab-paclitaxel 125 mg/m² (D1, D8, q3w) and S-1 (40 mg BID for body surface area < 1.25 m²; 50 mg BID for body surface area of 1.25-1.5 m²; and 60 mg BID for body surface area >1.5 m²; D1-14, q3w)
  Interventions: Drug: S1 or Gemcitabine
- Gem/nab (Active Comparator): Nab-paclitaxel 125 mg/m² (D1, D8, q3w) and Gemcitabine 1000 mg/m² (D1, D8, q3w)
  Interventions: Drug: S1 or Gemcitabine

INTERVENTIONS:
Drug: S1 or Gemcitabine — Gemcitabine 1000 mg/m² (D1, D8, q3w) and S-1 (40 mg BID for body surface area < 1.25 m²; 50 mg BID for body surface area of 1.25-1.5 m²; and 60 mg BID for body surface area >1.5 m²; D1-14, q3w)

SUMMARY:
A randomized multi-center phase II trial of nab-paclitaxel in combination with gemcitabine verus S1 with gemcitabine as first-Line treatment for locally advanced or metastatic pancreatic cancer

DETAILED DESCRIPTION:
A Phase II, open-label randomized, multicenter trial to compare nab-paclitaxel in combination with gemcitabine verus S1 with gemcitabine with respect to overall survival, objective tumor response rate and Progression Free Survival (PFS) in patients diagnosed with locally advanced or metastatic adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of pancreatic adenocarcinoma
* Distant metastatic or unresctable locally advanced diseases
* CTScan (or MRI if scanner contraindicated) completed within 3 weeks of the start of treatment
* At least one lesion measurable by RECIST v1.1 criteria
* Life expectancy> 3 months
* No previous chemotherapy (adjuvant chemotherapy with gemcitabine authorised if administered more than 6 months prior to inclusion)
* No previous radiotherapy (unless at least one measurable target lesion outside the irradiation zone)
* Pain must be monitored before inclusion
* 18 years < age < 70
* Performance status: 0-1
* ANC ≥ 1500/mm3, platelets ≥ 100 000/mm3, haemoglobin ≥ 9 g/dL
* ASAT (SGOT), ALAT (SGPT) ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases found
* Bilirubin ≤ 1.5 x ULN (patients drained by retrograde technique are includable),
* creatinine < 120 μmol/L, or MDRD creatinine clearance > 60 mL/min
* Patient information and signature of informed consent

Exclusion Criteria:

* Concurrent other effective treatment (including radiotherapy)
* Resectable patients
* Allergy history to other drugs in the same class patients with pregnancy or lactation
* Known severe internal medical diseases
* Abnormal heart function or relevant history of myocardial infarction and severe arrhythmia
* Immunocompromised patients, such as HIV positive
* Uncontrollable mental illness
* Other conditions the researchers considered ineligible for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 month
  progression-free survival

SECONDARY OUTCOMES:
OS | 1 year
  overall survival
ORR | 6 month
  objective response rate
DCR | 6 month
  CR+PR+SD was defined as disease control rate (DCR)
Safety profile :Adverse events of nab-Paclitaxel plus S-1 | 1 year
  Adverse events of nab-Paclitaxel plus S-1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Result] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081
- [Result] Xu Y, Guo X, Fan Y, Wang D, Wu W, Wu L, Liu T, Xu B, Feng Y, Wang Y, Lou W, Zhou Y. Efficacy and safety comparison of nabpaclitaxel plus S-1 and gemcitabine plus S-1 as first-line chemotherapy for metastatic pancreatic cancer. Jpn J Clin Oncol. 2018 Jun 1;48(6):535-541. doi: 10.1093/jjco/hyy063. PMID 29718363